CLINICAL TRIAL: NCT03788564
Title: The Association of Cardiac Ion Channel Related Gene Polymorphism and Prolonged QTc Interval After Endotracheal Intubation
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2017-0727
Record Dates: First submitted 2018-12-25; First posted 2018-12-27 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Emergence Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The QTc interval is affected by heart rate, medications and changes in the autonomic nervous system. The endotracheal laryngoscopy, the necessary step during general anesthesia, prolongs QTc interval. Changes in the flow of ion currents could result from the genetic variation of myocardial ion channels by gene polymorphism. This study is to investigate the association of cardiac ion channel related gene polymorphism and prolonged QTc interval after endotracheal intubation in adult patients.

ELIGIBILITY:
Inclusion Criteria:

1. 20-65 years old
2. scheduled for general anesthesia requiring direct laryngoscopy

Exclusion Criteria:

1. Patients taking antihypertensive medication (beta-blocker, CCB)
2. patients taking other medications known to affect QTc interval
3. Patients with abnormal ECG and prolonged QTc (>500 msec)
4. Diabetes, liver disease, kidney disease, heart failure, congenital heart disease
5. Severe electrolyte imbalance
6. illiterate, foreigners who cannot understand the consent form

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 20-65 years old, scheduled for general anesthesia requiring direct laryngoscopy
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2017-09-24 (Actual); Primary Completion 2020-05-03 (Actual); Study Completion 2020-05-03 (Actual)

PRIMARY OUTCOMES:
QTc interval | Before anesthesia, Before laryngoscopy, Right after laryngoscopy, 5 minutes after laryngoscopy
  QTc interval prolongs followed by laryngoscopy due to changes in the autonomic nervous system. The restoration of the prolonged QTc could also be affected by the balance of autonomic nervous system or changes in the related cardiac ion channels.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea